CLINICAL TRIAL: NCT00987571
Title: Carpal Tunnel Syndrome: Case Reports and Analysis - Ultrasound Imaging and Pathomechanics of Median Nerve Compression
Status: Completed | Type: Observational
Sponsor: EMG Labs of Arizona Arthritis & Rheumatology Associates (Other)
Responsible Party: Benjamin M. Sucher, D.O./Medical Director, EMG Labs of AARA
Other Study IDs: CTS-US Med N JAOA
Record Dates: First submitted 2009-09-29; First posted 2009-10-01 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; median nerve; ultrasound; electrodiagnosis; Normal subjects
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Carpal Tunnel patients: These patients have documented carpal tunnel syndrome
- Normal Subjects: These individuals have no carpal tunnel syndrome

SUMMARY:
Carpal tunnel syndrome is caused by compression of the median nerve at the wrist. The hypothesis is that ultrasound imaging can be used to visualize nerve compression in carpal tunnel patients during hand activity, and normal subjects will not demonstrate any nerve compression.

DETAILED DESCRIPTION:
Two patients with carpal tunnel syndrome underwent nerve testing to document that they had median nerve abnormality at the wrist. They subsequently had ultrasound imaging of the wrist at rest and during a stress test using hand activity. Two control subjects had nerve testing to prove that they had no nerve abnormality at the carpal tunnel. The carpal tunnel syndrome patients demonstrated nerve compression on the ultrasound images during the stress tests and the normal subjects showed no nerve compression.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have symptoms consistent with carpal tunnel syndrome and electrodiagnostic testing that demonstrates abnormal median nerve function at the wrist, consistent with carpal tunnel syndrome.
* Normal subjects must have no upper limb symptoms to support carpal tunnel syndrome and normal nerve testing.

Exclusion Criteria:

* Patients excluded if nerve testing was not consistent with carpal tunnel syndrome.
* Normals excluded if nerve testing demonstrated any median nerve abnormality.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with upper extremity symptoms of pain, numbness, and tingling; Adult subjects with no upper extremity pain, numbness, or tingling
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Median nerve compressive narrowing on ultrasound imaging in carpal tunnel syndrome patients | 5 months

SECONDARY OUTCOMES:
No median nerve compressive narrowing in normal subjects | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Sucher, DO, Principal Investigator — EMG Labs of AARA